CLINICAL TRIAL: NCT04125043
Title: Sensitivity and Specificity of the Red Reflex Test for Detecting Anterior and Posterior Segment Ophthalmic Pathology in the Pediatric Population
Brief Title: Accuracy of the Red Reflex Test in the Pediatric Population
Status: Completed | Type: Observational
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, William Madigan, Chief, Division of Ophtamology, Children's National Research Institute
Other Study IDs: Pro00011173
Record Dates: First submitted 2019-10-10; First posted 2019-10-14 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Abnormal Vitreous Humor Morphology; Abnormal Choroid Morphology; Optic Nerve Diseases; Retinal Disease; Retinal Hemorrhage
Keywords: Red reflex; Posterior ocular abnormalities
MeSH Terms: conditions — Optic Nerve Diseases; Retinal Diseases; Retinal Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RRT Group: Pediatric patients undergoing ocular screening tests
  Interventions: Diagnostic Test: Direct ophthalmoscope

INTERVENTIONS:
Diagnostic Test: Direct ophthalmoscope — Red reflex test

SUMMARY:
This study is designed to investigate the sensitivity and specificity of the Red Reflex Test (RRT), with and without dilation, for early detection of ocular abnormalities in children and newborns. The RRT functions by shining a light from an ophthalmoscope into a participant's eye and noting the presence or absence of a red glow. Despite its use in pediatric clinics for years, this test at times fails to detect significant ocular diseases, especially located in the back of the eye, threatening visual development in this population. Therefore, the investigators aim to quantify the utility of this test as a tool for screening by comparing these findings on RRT with those of retinal photography.

The investigators hypothesize that the sensitivity and specificity of the RRT will be sufficient for detecting anterior segment pathology but will be insufficient for detecting posterior segment pathology with or without dilation.

DETAILED DESCRIPTION:
Pediatric patients will be recruited through clinical practice at the designated study sites. Participants with known anterior segment or posterior segment pathology will be eligible for inclusion. Patients who have a history of disease, treatments and/or surgical procedures affecting the ability for normal pupillary reaction are excluded. An equal number of age matched participants with a normal anterior and posterior segment exam will be recruited from routine outpatient ophthalmology clinic appointments. Informed consent will be obtained and will include an option to be considered for medical photography. Participants may opt out of photography and still be included in the study. For Spanish speaking participants, an interpreter will be used for study recruitment and informed consent. A Spanish informed consent (developed by a Spanish medical translator from our English written consent) will be provided. Current estimated number of subjects required for the study is 200 total including 100 controls. Patient charts will be accessed from date of birth to patient's current age using either Cerner or Epic depending on the study site location. Examiners will include ophthalmology residents with one completed year of ophthalmology training. They will be blinded to participants' ophthalmologic history.

Pupil size will be recorded under ambient lighting conditions and the red reflex test (RRT) performed at 18 cm using a direct ophthalmoscope (Welch Allyn 11710 or similar). Each eye will then be inspected individually at 1 cm. Examiner description of the pupillary reflex in terms of color, brightness, and the presence or absence of potential anterior/posterior segment abnormality will be recorded using a standardized survey tool. The exam room lights will then be turned off and the pupils examined again with the direct ophthalmoscope according to the standard RRT procedure and results recorded.

Next, pharmacological dilation will be achieved according to standard practices. For all patients, one drop of proparacaine hydrochloride ophthalmic solution will be instilled in each eye to achieve anesthesia. For patients under 1 year old, one drop of Cyclomydril will then be instilled in each eye and followed second drop in each eye 5 minutes later. For children over 1 year of age, pharmacologic dilation will be achieved with 1 drop of Cyclopentolate 1% and 1 drop of Phenylephrine 2.5% in each eye. The RRT will be repeated by the same examiner, including the lights on and lights off portions of the exam, and the results recorded.

Subjects will be de-identified and results will be stored on a password protected Children's National Hospital computer and pertinent statistical analyses will be perform to asses our hypothesis. All statistical tests will be performed at the 5% level of significance unless otherwise stated.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients recruited in clinical practice with known anterior or posterior segment pathology as well as patients without anterior or posterior segment pathology

Exclusion Criteria:

* Patients who have a history of disease, treatments and/or surgical procedures affecting the ability for normal pupillary reaction

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pediatric patients under 18 years old recruited in clinical practice with known anterior or posterior segment pathology as well as patients without anterior or posterior segment pathology.
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity and Specificity of RRT | 1 year
  sensitivity and specificity of the RRT in detecting anterior segment pathology, as well as the sensitivity and specificity of the RRT in detecting posterior segment pathology

SECONDARY OUTCOMES:
Sensitivity and Specificity of RRT with Dilation | 1 year
  the sensitivity and specificity of the RRT in detecting anterior segment or posterior segmented pathology following pharmacologic dilation

CONTACTS AND LOCATIONS:
Overall Officials: William P Madigan, MD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-10-21): https://cdn.clinicaltrials.gov/large-docs/43/NCT04125043/Prot_SAP_ICF_001.pdf